CLINICAL TRIAL: NCT01227057
Title: Treatment of Late Life Compulsive Hoarding
Brief Title: Hoarding Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSRD-068-10S
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Results first posted 2016-06-03 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Compulsive Hoarding
Keywords: exposure therapy; case management; older adults; cognitive rehabilitation
MeSH Terms: interventions — Cognitive Training; Implosive Therapy; Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Cognitive Rehabilitation (Experimental): Cognitive rehabilitation and exposure therapy for hoarding
  Interventions: Behavioral: Cognitive Rehabilitation and Exposure Therapy for Compulsive Hoarding
- Arm 2: Case Management (Active Comparator): Case management
  Interventions: Behavioral: Case Management

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation and Exposure Therapy for Compulsive Hoarding — The intervention includes cognitive remediation for deficits in executive functioning and exposure therapy for discarding/acquiring.
  Arms: Arm 1: Cognitive Rehabilitation
Behavioral: Case Management — Case management
  Arms: Arm 2: Case Management

SUMMARY:
The purpose of this investigation is to examine treatment outcome of a new intervention for hoarding in older adults compared to standard case management for hoarding. The new intervention combines exposure therapy and cognitive remediation.

DETAILED DESCRIPTION:
Research has shown that hoarding disorder (HD) is debilitating chronic and progressive condition that has significant public health implications. Older adults represent the largest group of HD suffers due to increasing severity with age. Often, Veterans with HD are seen in the VA system and the status of their hoarding is never assessed. Providers are treating patients for other health and social service issues yet missing an important source of disability and distress. This insidious, often undetected condition leads to greater medical and social disability and is costly to the VA system as patients continue to decompensate. When HD is even detected, patients in the VA receive indefinite case management and inadequate treatment. The cases the investigators know about have caused significant financial burden to the investigators' system. Most importantly, HD causes significant impairment and poor quality of life for the Veterans, particularly older Veterans. Unfortunately, the investigators know nothing about how to treat late life HD. Nor do the investigators know how neurocognitive features impact treatment response, which the investigators strongly suspect influence treatment outcome. HD is a potentially treatable source of disability in the VA system - one that the VA must research and treat. This study represents the first randomized controlled trial of a novel intervention for the treatment of HD in older Veterans. The main objective of this proposal is to further refine and test a new treatment for hoarding in older Veterans (age 60-85) which will be accomplished through a series of treatment development phases (case series, open labeled trial) and a randomized controlled trial. The new treatment (Cognitive Remediation and Exposure Therapy for hoarding; CogRET) is hypothesis driven and based on late life anxiety literature, consultation with mentors, results of the pilot study using a standard cognitive-behavioral intervention, and several case series that will be completed prior to the start of the Career Development Award (CDA). The first draft of CogRET is complete and is currently being used with several case studies. The research and training plan is divided into 5 phases; 1) training and preparation 2) training, further case studies using CogRET, further modification of CogRET 3)training, open label trial of CogRET, further modification of CogRET 4) randomized controlled trial and 5) presenting, publishing, dissemination of results and submission of a VA Merit grant. Primary hypotheses include 1) when randomized to CogRET, older Veterans with HD will show significant decreases in acquisition, difficulty discarding, and excessive clutter compared to those randomized to case management and 2) executive functioning (EF) is a significant moderator of treatment response. Other mediators and moderates of treatment response (psychiatric, medical, demographic, etc.) will be explored.

ELIGIBILITY:
Inclusion Criteria:

Participants must be between the ages of 60 - 85 years old and meet clinical criteria for Compulsive Hoarding (CH) developed by the Steketee and Frost (2000) research group. These criteria include:

* significant amount of clutter in active living spaces
* the urge to collect, buy, or acquire things
* an extreme reluctance to part with items
* clutter accumulation that causes distress or interferes with functioning
* symptom duration of at least 6 months
* the reluctance to part with items is not accounted for by other psychiatric conditions.

To be enrolled, patients must have:

* a score of 20 or greater on the University of California, Los Angeles Hoarding Severity Scale (UHSS)
* 40 or greater on the Savings Inventory-Revised (SI-R)
* severity rating of 4 or higher on the Anxiety Disorders Interview Schedule (ADIS-IV) rating scales for clutter and difficulty discarding
* and diagnosis confirmed at a consensus conference including at least two licensed professionals with expertise in CH (myself and at least one mentor).

Exclusion Criteria:

* Individuals with moderate to severe cognitive deficits (scores below 23 on the MMSE) will be excluded.
* Prospective participants must not have active substance abuse problems.
* Participants will also be excluded if they are currently in other forms of psychotherapy.
* Participants must have no change in any psychotropic medications for at least three months prior to the initial assessment.
* Patients with current psychosis or mania will be excluded.
* Mood and anxiety disorders are permitted as long as compulsive hoarding is the primary diagnosis.
* Participants will are not eligible if they have active suicidal ideation, those participants will be given immediate medical or mental health attention.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine R Ayers, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

REFERENCES:
- [Derived] Ayers CR, Dozier ME, Twamley EW, Saxena S, Granholm E, Mayes TL, Wetherell JL. Cognitive Rehabilitation and Exposure/Sorting Therapy (CREST) for Hoarding Disorder in Older Adults: A Randomized Clinical Trial. J Clin Psychiatry. 2018 Mar/Apr;79(2):16m11072. doi: 10.4088/JCP.16m11072. PMID 28541646
- See also: Click here for more information about this study: Treatment of Late Life Compulsive Hoarding — http://ayerslab.wordpress.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Cognitive Rehabilitation | Arm 2: Case Management
Started | 31 | 27
Completed | 25 | 19
Not Completed | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Cognitive Rehabilitation | Arm 2: Case Management | Total
Number analyzed (Participants) | 31 | 27 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.35 (6.49) | 64.19 (5.35) | 66.95 (6.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 17 | 41
  Male | 7 | 10 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 27 | 24 | 51
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 31 | 27 | 58
Saving Inventory Revised [Mean (Standard Deviation); unit: units on a scale] — Total score is 0-92, with higher scores indicating worse hoarding severity.
  units on a scale | 57.35 (10.23) | 59.48 (14.01) | 58.34 (12.08)
Clutter Image Rating [Mean (Standard Deviation); unit: units on a scale] — Mean score is 1-9, with higher scores indicating worse clutter severity.
  units on a scale | 4.15 (1.71) | 4.33 (2.11) | 4.24 (1.89)
University of California, Los Angeles Hoarding Severity Scale [Mean (Standard Deviation); unit: units on a scale] — Total score is 0-40, with higher scores indicating worse hoarding severity.
  units on a scale | 26.35 (5.31) | 28.85 (5.82) | 27.52 (5.65)
Activities of Daily Living - Hoarding [Mean (Standard Deviation); unit: units on a scale] — Mean score is 1-75, with higher scores indicating worse impairment due to hoarding.
  units on a scale | 30.85 (9.3) | 31.90 (13.53) | 31.31 (11.23)
Hospital Anxiety and Depression [Mean (Standard Deviation); unit: units on a scale] — Total score for each subscale is 0-21, with higher scores indicating worse anxiety or depression severity.
  units on a scale
    Hospital Anxiety and Depression - Anxiety | 9.06 (4.39) | 10.15 (3.41) | 9.56 (3.98)
    Hospital Anxiety and Depression - Depression | 7.13 (3.23) | 8.56 (4.97) | 7.79 (4.16)
Clinician Global Improvement - Severity scale [Mean (Standard Deviation); unit: units on a scale] — Total score is 1-7, with higher scores indicating worse severity of mental illness.
  units on a scale | 3.67 (.92) | 3.96 (1.19) | 3.81 (1.06)

OUTCOME MEASURES:

1. Primary Outcome: Hoarding Symptom Severity as Measured by the Saving Inventory-Revised (SI-R) at 6 Months
Description: Hoarding symptom severity (primary outcome) will be measured using the Savings Inventory-Revised (SI-R), a 23-item self-report measure used to assess common hoarding symptoms. Subtests include excessive clutter, compulsive acquisition, and difficulty discarding. The SI-R has demonstrated good internal consistency, divergent validity, concurrent validity, divergent validity, test-retest reliability in clinical samples with hoarding. The total score will be used for analyses. The range of the total score is 0-92, with higher scores indicating worse hoarding severity.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Cognitive Rehabilitation | Arm 2: Case Management
Number analyzed (Participants) | 25 | 19
units on a scale | 35.44 (15.48) | 44.68 (13.29)
Statistical Analysis 1: Comparison: Arm 1: Cognitive Rehabilitation vs Arm 2: Case Management; Linear mixed models with random intercepts were used to evaluate the change in primary and secondary outcome variables over time, the effect of group, the effect of treatment, and the treatment group by time interaction, both for the treatment phase (0-6 months) and follow up phase (6-12 months). All analyses (0-6 months) were conducted first using observed data only (i.e., completer analysis) and then using an intent to treat (ITT) sample; Test type: Non-Inferiority or Equivalence — Power calculations were based on the SI-R using effect size estimates from a previous trial comparing individual CBT with a Wait List (WL) control (Steketee2010). In this study, the effect size of Cognitive Behavioral Therapy (CBT) relative to WL was d = 2.21 on the SI-R. Accounting for a smaller effect size due to having an active control condition, we expected to have 80% power to detect a large (d = .80) effect size. The sample assessed for eligibility (n = 67) was 99% of this target; p = .029, Mixed Models Analysis — P value is for the group x time interaction; Adjusted for age, years of education, and presence of co-morbid obsessive-compulsive disorder due to group differences at baseline

2. Secondary Outcome: The Activities of Daily Living in Hoarding (ADL-H)
Description: The Activities of Daily Living in Hoarding (ADL-H) was used to assess functional impairment. Higher scores represent increased impairment. Mean score is 1-75, with higher scores indicating worse impairment due to hoarding.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Cognitive Rehabilitation | Arm 2: Case Management
Number analyzed (Participants) | 25 | 19
units on a scale | 21.09 (6.67) | 27.81 (14.29)
Statistical Analysis 1: Comparison: Arm 1: Cognitive Rehabilitation vs Arm 2: Case Management; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .04, Mixed Models Analysis — P value is for the group x time interaction; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Executive Functioning as Measured by the Delis Kaplan Executive Functioning System (D-KEFS) at 6 Months
Description: The D-KEFS Trail Making Test Condition 4: Number-Letter Switching Scaled Score was used to assess executive functioning. Scaled scores range from 1-19. Higher scores represent less impairment.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Cognitive Rehabilitation | Arm 2: Case Management
Number analyzed (Participants) | 25 | 19
units on a scale | 10.8 (3.67) | 10.8 (3.11)
Statistical Analysis 1: Comparison: Arm 1: Cognitive Rehabilitation vs Arm 2: Case Management; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .1, ANOVA — P value is for the group x time interaction

ADVERSE EVENTS:
Arm/Group | Arm 1: Cognitive Rehabilitation | Arm 2: Case Management
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/27
Other Adverse Events (participants affected / at risk) | 0/31 | 0/27

LIMITATIONS AND CAVEATS:
The study was under-powered to fully detect the differences between CREST and Case Management.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes